CLINICAL TRIAL: NCT01072565
Title: Optimization of SMBG Employing Modal Day Analysis: Examining Clinical Decision-making Processes Using Blinded FreeStyle Navigator Continuous Glucose Monitoring System (CGM)
Brief Title: Modal Day Analysis of Self Monitoring Blood Glucose Versus Continuous Glucose Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 03914-09-C
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; A1c; Continuous Glucose Monitoring; Blood Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMBG Only (Active Comparator): You will measure your blood glucose 4 times daily by finger sticks using a blood glucose meter and you will also wear a CGM device. The CGM measurements will be blinded (neither you nor the study doctor will be able to see the CGM measurements until your final study visit). Only your SMBG measurements will be considered to help manage your diabetes. Your medications will be changed or adjusted based on your HbA1c and/or glucose readings with a goal to achieve an HbA1c level of less than 7%.
  Interventions: Other: SMBG to guide clinical decisions
- SMBG and CGM (Active Comparator): You will measure your blood glucose 4 times daily by finger sticks using a blood glucose meter and you will also wear a CGM device. The CGM measurements will be downloaded at each study visit and will be considered along with your SMBG measurements to help manage your diabetes. Your medications will be changed or adjusted based on your HbA1c and/or glucose readings with a goal to achieve an HbA1c level of 7%.
  Interventions: Other: SMBG and CGM

INTERVENTIONS:
Other: SMBG to guide clinical decisions — The investigator will base clinical decisions on A1c and modal day analysis of SMBG.
  Arms: SMBG Only
Other: SMBG and CGM — The investigator will base clinical decisions on A1c, modal day analysis of SMBG and CGM data.
  Arms: SMBG and CGM

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Self Monitoring of Blood Glucose (SMBG) for clinical decisions related to the management of type 2 diabetes and to determine the benefit of using Continuous Glucose Monitoring (CGM) for clinical diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 and ≤75 years of age
* Clinical diagnosis of diabetes
* Diabetes duration ≥ 1 year
* HbA1c ≥7.2%
* Diabetes can be treated with any therapy including medical nutrition therapy alone and any pharmaceutical therapy

Exclusion Criteria:

* Taken prednisone or cortisone medications in the previous 30 days
* Currently pregnant or planning pregnancy during the study period
* Presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study
* Unable to follow the study protocol
* Unable to speak, read and write in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of SMBG for clinical decisions related to the management of type 2 diabetes. | Three, six and nine months.

SECONDARY OUTCOMES:
Determine the incremental benefit of CGM for clinical decision-making. | Three, six and nine months.

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Mazze, PhD, Principal Investigator — International Diabetes Center at Park Nicollet; Elinor S Strock, APRN, BC, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States